CLINICAL TRIAL: NCT04025840
Title: Effect of Perioperative Epidural Block and Dexamethasone on Outcome of Patients Undergoing Pancreatic Cancer Surgery: a 2×2 Factorial Randomized Controlled Trial
Brief Title: Perioperative Epidural Block and Dexamethasone in Pancreatic Cancer Surgery
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Chairman, Department of Anaesthesiology and Critical Care Medicine, Peking University First Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019-99
Record Dates: First submitted 2019-07-16; First posted 2019-07-19 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Cancer; Surgery; Epidural Block; Dexamethasone; Overall Survival
Keywords: Pancreatic cancer; Radical resection; Epidural block; Dexamethasone; Overall survival
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Anesthesia, Epidural; Analgesia; Dexamethasone; Glucocorticoids

STUDY DESIGN:
Intervention Model Description: 2×2 factorial trial
Who Masked: Outcomes Assessor
Masking Description: For dexamethasone administration, all the participants, care providers, investigators, and outcomes assessors are masked. For epidural block, outcome assessors are masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Patients in this group receive general anesthesia, without epidural block and perioperative dexamethasone. Patient-controlled intravenous analgesia is provided after surgery.
- Epidural block (Experimental): Patients in this group receive combined epidural-general anesthesia (0.375% ropivacaine for epidural block), without perioperative dexamethasone. Patient-controlled epidural analgesia is provided after surgery.
  Interventions: Other: Epidural block
- Dexamethasone (Experimental): Patients in this group receive dexamethasone (10 mg) before anesthesia induction and general anesthesia, without epidural block. Patient-controlled intravenous analgesia is provided after surgery.
  Interventions: Drug: Dexamethasone
- Epidural block+Dexamethasone (Experimental): Patients this group receive dexamethasone (10 mg) before anesthesia induction and combined epidural-general anesthesia (0.375% ropivacaine for epidural block). Patient-controlled epidural analgesia is provided after surgery.
  Interventions: Other: Epidural block; Drug: Dexamethasone

INTERVENTIONS:
Other: Epidural block — Epidural block (with 0.375% ropivacaine) is performed during surgery. Patient-controlled epidural analgesia (with a mixture of 0.12% ropivacaine and 0.5 microgram/ml sufentanyl) is provided after surgery.
  Other Names: Epidural anesthesia/analgesia
  Arms: Epidural block; Epidural block+Dexamethasone
Drug: Dexamethasone — Dexamethasone (10 mg) is administered intravenously before anesthesia induction.
  Other Names: Glucocorticoids
  Arms: Dexamethasone; Epidural block+Dexamethasone

SUMMARY:
Pancreatic cancer remains a devastating disease with an average 5-year survival rate of about 3-5%. Previous retrospective studies showed that perioperative epidural block and/or dexamethasone are associated with improved outcome after cancer surgery. This randomized trial aims to investigate the effect of perioperative epidural block and/or dexamethasone on long-term survival in patients following pancreatic cancer surgery.

DETAILED DESCRIPTION:
Pancreatic cancer is the fourth leading cause of cancer-related death in the world, and is estimated to become the second one in 2030. For patients with resectable pancreatic cancer, radical surgery is the first-line therapy. However, the clinical outcomes remain poor even after radical resection, as the incidence of postoperative morbidity is up to 50% and the 5-year survival rate remains below 30%.

For patients undergoing major intraabdominal surgery, epidural block may provide advantages by blocking the afferent nociceptive stimuli, providing better pain relief, decreasing opioid consumption, and alleviating stress response. These effects may be helpful in preserving immune function. Some retrospective studies showed that epidural block is associated with delayed cancer recurrence/metastasis and improved survival after cancer surgery.

Low-dose dexamethasone is frequently used to prevent postoperative nausea and vomiting. Recent evidences from retrospective studies suggest that perioperative dexamethasone may also affect long-term outcome after cancer surgery. For example, in patients undergoing lung cancer surgery, intraoperative dexamethasone is associated with improved recurrence-free and overall survival. Similar results are also reported in patients after pancreatic cancer surgery.

The investigators hypothesize that perioperative epidural block and dexamethasone may improve survival in patients after radical pancreatic surgery. The purpose of this study is to investigate whether perioperative epidural block and/or dexamethasone can improve 2-year survival in patients after pancreatic cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥45 and <90 years;
2. Clinically diagnosed as resectable or possibly resectable pancreatic cancer and scheduled to undergo radical surgery;
3. Agreed to receive epidural block and postoperative patient-controlled analgesia;
4. Agreed to participate in the study and provided written informed consent.

Exclusion Criteria:

1. Clinical evidence of unresectable pancreatic cancer or plan to undergo biopsy;
2. Previous surgery for pancreatic cancer, scheduled to undergo resurgery for recurrence or metastasis;
3. Complicated with primary malignant tumor in other organ(s), either previously or at present;
4. Complicated with autoimmune diseases, receiving either glucocorticoids or other immunosuppressants before surgery;
5. Unable to complete preoperative evaluation due to severe dementia, language barrier, coma, or end-stage diseases;
6. Severe hepatic dysfunction (Child-Pugh C), severe renal insufficiency (serum creatinine >442 µmol/L or requirement of renal replacement therapy), or American Society of Anesthesiologists classification ≥V；
7. Contradictions to epidural anesthesia, including spinal malformation, history of spinal surgery, coagulation disorder, suspected infection at the site of puncture, or severe low back pain;
8. Other conditions that are considered unsuitable for study participation;
9. Refused to participate in the study.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
2-year overall survival | Up to 2 years after surgery.
  2-year overall survival

SECONDARY OUTCOMES:
Postoperative gastrointestinal complications. | Up to 30 days after surgery.
  Rate of postoperative gastrointestinal complications.
Overall postoperative complications. | Up to 30 days after surgery.
  Rate of overall postoperative complications.
Length of stay in hospital after surgery. | Up to 30 days after surgery.
  Length of stay in hospital after surgery.
All-cause 30-day mortality. | Up to 30 days after surgery.
  Rate of all-cause 30-day mortality.
Quality of life in 1- and 2-year survivors. | At the end of the first and second year after surgery.
  Quality of life is assessed with the European Organization for Research and Treatment of Cancer Quality of Life Questionaire (EORTC QLQ)-PAN26. It is a 26-item questionnaire that evaluates 9 symptoms and 5 emotional difficulties related to pancreatic cancer. Each item is scaled 0-100. High scores indicate worse symptoms and poorer quality of life.
Hospital readmission within 2 years after surgery. | Up to 2 years after surgery.
  Rate of hospital readmission within 2 years after surgery.
2-year progression-free survival | Up to 2 years after surgery.
  Cancer progression is evaluated according to the Response Evaluation Criteria in Solid Tumors (RECIST) guideline version 1.1.

OTHER OUTCOMES:
Subjective sleep quality: Numeric Rating Scale | Between 8-10 am on the first, second, and third days after surgery.
  Subjective sleep quality is assessed with a Numeric Rating Scale (NRS, an 11-point scale where 0 indicates the best sleep and 10 the worst sleep).
Pain severity (at rest and with movement): Numeric Rating Scale | Between 8-10 am on the first, second, and third days after surgery.
  Pain severity is assessed with a Numeric Rating Scale (NRS, an 11-point scale where 0 indicates no pain and 10 the worst pain).
Time to ambulation after surgery. | Up to 30 days after surgery.
  Time to ambulation after surgery.
Time to oral intake after surgery. | Up to 30 days after surgery.
  Time to oral intake after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2018. CA Cancer J Clin. 2018 Jan;68(1):7-30. doi: 10.3322/caac.21442. Epub 2018 Jan 4. PMID 29313949
- [Background] Rahib L, Smith BD, Aizenberg R, Rosenzweig AB, Fleshman JM, Matrisian LM. Projecting cancer incidence and deaths to 2030: the unexpected burden of thyroid, liver, and pancreas cancers in the United States. Cancer Res. 2014 Jun 1;74(11):2913-21. doi: 10.1158/0008-5472.CAN-14-0155. PMID 24840647
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Chen W, Sun K, Zheng R, Zeng H, Zhang S, Xia C, Yang Z, Li H, Zou X, He J. Cancer incidence and mortality in China, 2014. Chin J Cancer Res. 2018 Feb;30(1):1-12. doi: 10.21147/j.issn.1000-9604.2018.01.01. PMID 29545714
- [Background] Kamisawa T, Wood LD, Itoi T, Takaori K. Pancreatic cancer. Lancet. 2016 Jul 2;388(10039):73-85. doi: 10.1016/S0140-6736(16)00141-0. Epub 2016 Jan 30. PMID 26830752
- [Background] Yeo CJ, Cameron JL. Prognostic factors in ductal pancreatic cancer. Langenbecks Arch Surg. 1998 Apr;383(2):129-33. doi: 10.1007/s004230050104. PMID 9641885
- [Background] Winter JM, Cameron JL, Campbell KA, Arnold MA, Chang DC, Coleman J, Hodgin MB, Sauter PK, Hruban RH, Riall TS, Schulick RD, Choti MA, Lillemoe KD, Yeo CJ. 1423 pancreaticoduodenectomies for pancreatic cancer: A single-institution experience. J Gastrointest Surg. 2006 Nov;10(9):1199-210; discussion 1210-1. doi: 10.1016/j.gassur.2006.08.018. PMID 17114007
- [Background] Heerkens HD, Tseng DS, Lips IM, van Santvoort HC, Vriens MR, Hagendoorn J, Meijer GJ, Borel Rinkes IH, van Vulpen M, Molenaar IQ. Health-related quality of life after pancreatic resection for malignancy. Br J Surg. 2016 Feb;103(3):257-66. doi: 10.1002/bjs.10032. Epub 2015 Nov 19. PMID 26785646
- [Background] Ohtsuka T, Yamaguchi K, Chijiiwa K, Kinukawa N, Tanaka M. Quality of life after pylorus-preserving pancreatoduodenectomy. Am J Surg. 2001 Sep;182(3):230-6. doi: 10.1016/s0002-9610(01)00709-7. PMID 11587683
- [Background] Conroy T, Bachet JB, Ayav A, Huguet F, Lambert A, Caramella C, Marechal R, Van Laethem JL, Ducreux M. Current standards and new innovative approaches for treatment of pancreatic cancer. Eur J Cancer. 2016 Apr;57:10-22. doi: 10.1016/j.ejca.2015.12.026. Epub 2016 Feb 4. PMID 26851397
- [Background] Chae BK, Lee HW, Sun K, Choi YH, Kim HM. The effect of combined epidural and light general anesthesia on stress hormones in open heart surgery patients. Surg Today. 1998;28(7):727-31. doi: 10.1007/BF02484619. PMID 9697266
- [Background] Popping DM, Elia N, Van Aken HK, Marret E, Schug SA, Kranke P, Wenk M, Tramer MR. Impact of epidural analgesia on mortality and morbidity after surgery: systematic review and meta-analysis of randomized controlled trials. Ann Surg. 2014 Jun;259(6):1056-67. doi: 10.1097/SLA.0000000000000237. PMID 24096762
- [Background] Guay J. The effect of neuraxial blocks on surgical blood loss and blood transfusion requirements: a meta-analysis. J Clin Anesth. 2006 Mar;18(2):124-8. doi: 10.1016/j.jclinane.2005.08.013. PMID 16563330
- [Background] Haughom BD, Schairer WW, Nwachukwu BU, Hellman MD, Levine BR. Does Neuraxial Anesthesia Decrease Transfusion Rates Following Total Hip Arthroplasty? J Arthroplasty. 2015 Sep;30(9 Suppl):116-20. doi: 10.1016/j.arth.2015.01.058. Epub 2015 Jun 3. PMID 26077150
- [Background] Waurick R, Van Aken H. Update in thoracic epidural anaesthesia. Best Pract Res Clin Anaesthesiol. 2005 Jun;19(2):201-13. doi: 10.1016/j.bpa.2004.12.001. PMID 15966493
- [Background] Biki B, Mascha E, Moriarty DC, Fitzpatrick JM, Sessler DI, Buggy DJ. Anesthetic technique for radical prostatectomy surgery affects cancer recurrence: a retrospective analysis. Anesthesiology. 2008 Aug;109(2):180-7. doi: 10.1097/ALN.0b013e31817f5b73. PMID 18648226
- [Background] Exadaktylos AK, Buggy DJ, Moriarty DC, Mascha E, Sessler DI. Can anesthetic technique for primary breast cancer surgery affect recurrence or metastasis? Anesthesiology. 2006 Oct;105(4):660-4. doi: 10.1097/00000542-200610000-00008. PMID 17006061
- [Background] Tsui BC, Rashiq S, Schopflocher D, Murtha A, Broemling S, Pillay J, Finucane BT. Epidural anesthesia and cancer recurrence rates after radical prostatectomy. Can J Anaesth. 2010 Feb;57(2):107-12. doi: 10.1007/s12630-009-9214-7. PMID 19911247
- [Background] Wuethrich PY, Hsu Schmitz SF, Kessler TM, Thalmann GN, Studer UE, Stueber F, Burkhard FC. Potential influence of the anesthetic technique used during open radical prostatectomy on prostate cancer-related outcome: a retrospective study. Anesthesiology. 2010 Sep;113(3):570-6. doi: 10.1097/ALN.0b013e3181e4f6ec. PMID 20683253
- [Background] Wang J, Guo W, Wu Q, Zhang R, Fang J. Impact of Combination Epidural and General Anesthesia on the Long-Term Survival of Gastric Cancer Patients: A Retrospective Study. Med Sci Monit. 2016 Jul 8;22:2379-85. doi: 10.12659/msm.899543. PMID 27386842
- [Background] Cummings KC 3rd, Xu F, Cummings LC, Cooper GS. A comparison of epidural analgesia and traditional pain management effects on survival and cancer recurrence after colectomy: a population-based study. Anesthesiology. 2012 Apr;116(4):797-806. doi: 10.1097/ALN.0b013e31824674f6. PMID 22273991
- [Background] Gottschalk A, Ford JG, Regelin CC, You J, Mascha EJ, Sessler DI, Durieux ME, Nemergut EC. Association between epidural analgesia and cancer recurrence after colorectal cancer surgery. Anesthesiology. 2010 Jul;113(1):27-34. doi: 10.1097/ALN.0b013e3181de6d0d. PMID 20508494
- [Background] Grandhi RK, Lee S, Abd-Elsayed A. The Relationship Between Regional Anesthesia and Cancer: A Metaanalysis. Ochsner J. 2017 Winter;17(4):345-361. PMID 29230120
- [Background] Perez-Gonzalez O, Cuellar-Guzman LF, Soliz J, Cata JP. Impact of Regional Anesthesia on Recurrence, Metastasis, and Immune Response in Breast Cancer Surgery: A Systematic Review of the Literature. Reg Anesth Pain Med. 2017 Nov/Dec;42(6):751-756. doi: 10.1097/AAP.0000000000000662. PMID 28953508
- [Background] Giles AJ, Hutchinson MND, Sonnemann HM, Jung J, Fecci PE, Ratnam NM, Zhang W, Song H, Bailey R, Davis D, Reid CM, Park DM, Gilbert MR. Dexamethasone-induced immunosuppression: mechanisms and implications for immunotherapy. J Immunother Cancer. 2018 Jun 11;6(1):51. doi: 10.1186/s40425-018-0371-5. PMID 29891009
- [Background] Kunicka JE, Talle MA, Denhardt GH, Brown M, Prince LA, Goldstein G. Immunosuppression by glucocorticoids: inhibition of production of multiple lymphokines by in vivo administration of dexamethasone. Cell Immunol. 1993 Jun;149(1):39-49. doi: 10.1006/cimm.1993.1134. PMID 8513511
- [Background] Yu HC, Luo YX, Peng H, Kang L, Huang MJ, Wang JP. Avoiding perioperative dexamethasone may improve the outcome of patients with rectal cancer. Eur J Surg Oncol. 2015 May;41(5):667-73. doi: 10.1016/j.ejso.2015.01.034. Epub 2015 Feb 19. PMID 25744813
- [Background] Singh PP, Lemanu DP, Taylor MH, Hill AG. Association between preoperative glucocorticoids and long-term survival and cancer recurrence after colectomy: follow-up analysis of a previous randomized controlled trial. Br J Anaesth. 2014 Jul;113 Suppl 1:i68-73. doi: 10.1093/bja/aet577. Epub 2014 Feb 27. PMID 24583820
- [Background] Huang WW, Zhu WZ, Mu DL, Ji XQ, Nie XL, Li XY, Wang DX, Ma D. Perioperative Management May Improve Long-term Survival in Patients After Lung Cancer Surgery: A Retrospective Cohort Study. Anesth Analg. 2018 May;126(5):1666-1674. doi: 10.1213/ANE.0000000000002886. PMID 29517574
- [Background] Sandini M, Ruscic KJ, Ferrone CR, Warshaw AL, Qadan M, Eikermann M, Lillemoe KD, Fernandez-Del Castillo C. Intraoperative Dexamethasone Decreases Infectious Complications After Pancreaticoduodenectomy and is Associated with Long-Term Survival in Pancreatic Cancer. Ann Surg Oncol. 2018 Dec;25(13):4020-4026. doi: 10.1245/s10434-018-6827-5. Epub 2018 Oct 8. PMID 30298316
- [Background] Call TR, Pace NL, Thorup DB, Maxfield D, Chortkoff B, Christensen J, Mulvihill SJ. Factors associated with improved survival after resection of pancreatic adenocarcinoma: a multivariable model. Anesthesiology. 2015 Feb;122(2):317-24. doi: 10.1097/ALN.0000000000000489. PMID 25305092
- [Background] Katayama H, Kurokawa Y, Nakamura K, Ito H, Kanemitsu Y, Masuda N, Tsubosa Y, Satoh T, Yokomizo A, Fukuda H, Sasako M. Extended Clavien-Dindo classification of surgical complications: Japan Clinical Oncology Group postoperative complications criteria. Surg Today. 2016 Jun;46(6):668-85. doi: 10.1007/s00595-015-1236-x. Epub 2015 Aug 20. PMID 26289837
- [Background] Fitzsimmons D, Johnson CD, George S, Payne S, Sandberg AA, Bassi C, Beger HG, Birk D, Buchler MW, Dervenis C, Fernandez Cruz L, Friess H, Grahm AL, Jeekel J, Laugier R, Meyer D, Singer MW, Tihanyi T. Development of a disease specific quality of life (QoL) questionnaire module to supplement the EORTC core cancer QoL questionnaire, the QLQ-C30 in patients with pancreatic cancer. EORTC Study Group on Quality of Life. Eur J Cancer. 1999 Jun;35(6):939-41. doi: 10.1016/s0959-8049(99)00047-7. PMID 10533475
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Wente MN, Bassi C, Dervenis C, Fingerhut A, Gouma DJ, Izbicki JR, Neoptolemos JP, Padbury RT, Sarr MG, Traverso LW, Yeo CJ, Buchler MW. Delayed gastric emptying (DGE) after pancreatic surgery: a suggested definition by the International Study Group of Pancreatic Surgery (ISGPS). Surgery. 2007 Nov;142(5):761-8. doi: 10.1016/j.surg.2007.05.005. PMID 17981197
- [Background] Bassi C, Dervenis C, Butturini G, Fingerhut A, Yeo C, Izbicki J, Neoptolemos J, Sarr M, Traverso W, Buchler M; International Study Group on Pancreatic Fistula Definition. Postoperative pancreatic fistula: an international study group (ISGPF) definition. Surgery. 2005 Jul;138(1):8-13. doi: 10.1016/j.surg.2005.05.001. PMID 16003309
- [Background] Koch M, Garden OJ, Padbury R, Rahbari NN, Adam R, Capussotti L, Fan ST, Yokoyama Y, Crawford M, Makuuchi M, Christophi C, Banting S, Brooke-Smith M, Usatoff V, Nagino M, Maddern G, Hugh TJ, Vauthey JN, Greig P, Rees M, Nimura Y, Figueras J, DeMatteo RP, Buchler MW, Weitz J. Bile leakage after hepatobiliary and pancreatic surgery: a definition and grading of severity by the International Study Group of Liver Surgery. Surgery. 2011 May;149(5):680-8. doi: 10.1016/j.surg.2010.12.002. Epub 2011 Feb 12. PMID 21316725